CLINICAL TRIAL: NCT03737474
Title: A Multi-center, Open-label Trial to Assess the Long-term Safety and Efficacy of Brexpiprazole as Adjunctive Therapy in Patients With Major Depressive Disorder
Brief Title: A Long-Term Study of Brexpiprazole in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-102-00059
Record Dates: First submitted 2018-07-29; First posted 2018-11-09 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brexpiprazole (Experimental): 2 mg/day (starting dose 1mg/day) of Brexpiprazole will be orally administered once daily
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — 2 mg/day (starting dose 1mg/day) of Brexpiprazole will be orally administered once daily

SUMMARY:
This trial is a 52-week study to assess the safety of long-term use of brexpiprazole as adjunctive therapy in combination with an antidepressant.

ELIGIBILITY:
Inclusion Criteria:

* Rollover subjects

  1. Outpatients
  2. Subjects who have completed the double-blind period of the double-blind trial and can commence the treatment period of this trial within 28 days from the completionof the double-blind period of the double-blind trial
  3. Subjects who have a level of comprehension sufficient to allow them to give written informed consent to all of the observation/examination/evaluation items specified in the protocol, and who can understand the contents of the trial
  4. Subjects with a DSM-5 classification-based diagnosis of "major depressive disorder, single episode" or "major depressive disorder, recurrent episode"
* New subjects

  1. Outpatients
  2. Male and female patients ≥ 65 years of age (at the time of informed consent)
  3. Subjects who have a level of comprehension sufficient to allow them to give written informed consent to all of the observation/examination/evaluation items specified in the protocol, and who can understand the contents of the trial
  4. Patients with a DSM-5 classification-based diagnosis of "major depressive disorder, single episode" or "major depressive disorder, recurrent episode" whose current episode has persisted for at least 8 weeks

Exclusion Criteria:

* Rollover subjects

  1. Female subjects who are pregnant or breastfeeding or who have positive pregnancy test (urine) results at baseline
  2. Sexually active male subjects or sexually active female subjects of childbearing potential, who will not agree to practice 2 different methods of birth control or to remain abstinent during the trial and for 30 days after the final IMP administration. For birth control, 2 of the following methods must be used: vasectomy, tubal ligation, vaginal diaphragm, intra-uterine contraceptive device (IUD), oral contraceptives, or condom with spermicide.
  3. Subjects who experience a change to the manic state in the antidepressant treatment period of the double-blind trial
  4. Subjects who are discovered to not meet the inclusion criteria or to fall under any of the exclusion criteria in the doubleblind trial
  5. Subjects who showed marked noncompliance with the IMP treatment in the double-blind trial (subjects whose IMP compliance rates are < 65% between prescribed visits)
* New subjects

  1. Sexually active male subjects who will not agree to practice 2different methods of birth control or to remain abstinent during the trial and for 30 days after the final IMP administration. For birth control, 2 of the following methods must be used: vasectomy, tubal ligation, vaginal diaphragm, intra-uterine contraceptive device (IUD), oral contraceptives, or condom with spermicide.
  2. Patients with a treatment history showing that all antidepressants (also including those not used for the current major depressive episode) cannot be tolerated
  3. Patients with a history of electroconvulsive therapy
  4. Patients with a diagnosis of any of the following diseases according to DSM-5

     1. Neurocognitive disorders
     2. Schizophrenia spectrum and other psychotic disorders
     3. Bipolar and related disorders
     4. Feeding and eating disorders
     5. Obsessive-compulsive disorder
     6. Panic disorder
     7. Posttraumatic stress disorder

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-04-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nanko-kokorono clinic, Shirakawa, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

REFERENCES:
- [Derived] Kato M, Shiosakai M, Kuwahara K, Iba K, Shimada Y, Saito M, Sekine D, Aoki K, Shiomi Y, Higuchi T. A Multicenter, Open-Label Study to Evaluate the Long-term Safety and Efficacy of Adjunctive Brexpiprazole 2 mg Daily in Japanese Patients with Major Depressive Disorder. CNS Drugs. 2024 Dec;38(12):1003-1016. doi: 10.1007/s40263-024-01124-w. Epub 2024 Oct 18. PMID 39424742

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 248 participants in Japan. Of the 248 subjects who were administered investigational medicinal product, the efficacy analysis set and the safety analysis set comprised 247 subjects (216 rollover subjects, 31 newly enrolled subjects) of the total brexpiprazole population.
Groups:
- New Subjects: Newly entering elderly patients with major depressive disorder, aged 65 and over. 2 mg/day (starting dose 1mg/day) of Brexpiprazole were orally administered once daily.
- Rollover Subjects: Participants who rolled over from, and received blinded brexpiprazole or placebo in the randomized, double-blind, placebo-controlled Phase 2/3 efficacy studies (331-102-00058); 2 mg/day (starting dose 1mg/day) of Brexpiprazole were orally administered once daily
Period: Overall Study
Arm/Group | New Subjects | Rollover Subjects
Started | 31 | 216
Completed | 6 | 132
Not Completed | 25 | 84
Not completed — Adverse Event | 18 | 48
Not completed — Lack of Efficacy | 1 | 3
Not completed — Protocol Violation | 0 | 8
Not completed — Withdrawal by Subject | 5 | 20
Not completed — Non-compliance With Study Drug | 0 | 1
Not completed — Physician Decision | 1 | 4

BASELINE CHARACTERISTICS:
Population: This trial was conducted in 248 participants in Japan. Of the 248 subjects who were administered investigational medicinal product, the efficacy analysis set and the safety analysis set comprised 247 subjects (216 rollover subjects, 31 newly enrolled subjects) of the total brexpiprazole population.
Groups:
- Total: Total of all reporting groups
Arm/Group | New Subjects | Rollover Subjects | Total
Number analyzed (Participants) | 31 | 216 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 216 | 216
  >=65 years | 31 | 0 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.3 (4.5) | 40.7 (10.3) | 44.4 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 83 | 101
  Male | 13 | 133 | 146
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 31 | 216 | 247
Region of Enrollment [Number; unit: participants]
  Japan | 31 | 216 | 247

OUTCOME MEASURES:

1. Primary Outcome: The Frequency of Subjects With Treatment-Emergent Adverse Events (TEAEs)
Description: A treatment-emergent adverse event (TEAE) was defined as an AE that started after start of investigational medicinal product (IMP) treatment.
Time Frame: From baseline to week 52
Population: The safety analysis set comprised subjects who have received at least 1 dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | New Subjects | Rollover Subjects
Number analyzed (Participants) | 31 | 216
percentage of participants | 96.8 | 93.1

2. Secondary Outcome: Mean Changes From Baseline in Montgomery Åsberg Depression Rating Scale(MADRS) Total Scores at Week 52(LOCF)
Description: The MADRS was a clinician-rated scale which evaluated the level of depression.The MADRS consists of 10 items assessed apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thought. Each item was scored from 0 to 6, with higher scores indicating worse condition. Summed subscales were combined to compute a total score. Total score ranges from 0 to 60, with higher scores indicating worse condition.
Time Frame: Baseline and Week 52(LOCF)
Population: The efficacy analysis set comprised subjects who have received at least 1 dose of the IMP, and from whom MADRS total scores have been obtained at baseline and at least 1 time point after initiation of the treatment.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | New Subjects | Rollover Subjects
Number analyzed (Participants) | 31 | 216
Units on a scale | -2.8 (10.4) | -4.9 (9.0)

3. Secondary Outcome: The Proportion of Subjects Who Score 1 or 2 on the Clinical Global Impression-Improvement(CGI-I) Scale at Week 52(LOCF)
Description: The CGI-I Scale was clinician-rated scale which assessed the total improvement of the patient's condition compared to that at baseline. Scores range from 0 to 7: 0 = Not assessed, 1= Very much improved, 2 = Much improved, 3= Minimally improved, 4= No change, 5= Minimally worse, 6= Much worse, 7= Very much worse. Higher scores indicate worse condition.
Time Frame: Baseline and Week 52 (LOCF)
Population: The efficacy analysis set comprised subjects who have received at least 1 dose of theIMP, and from whom MADRS total scores have been obtained at baseline and at least 1 time point after initiation of the treatment.
Measure: Number; unit: percentage of Participants
Arm/Group | New Subjects | Rollover Subjects
Number analyzed (Participants) | 31 | 216
percentage of Participants | 29.0 | 37.0

4. Secondary Outcome: Mean Changes From Baseline in Clinical Global Impression-Severity of Illness(CGI-S) at Week 52(LOCF)
Description: The CGI-S Scale was a clinician-rated scale which assessed how mentally ill the patient is at the time. Scores range from 0 to 7: 0 = Not assessed, 1= Normal, not at all ill, 2 =Borderline mentally ill, 3= Mildly ill, 4= Moderately ill, 5= Markedly ill, 6= Severely ill, 7= Among the most extremely ill patients. Higher scores indicate worse condition.
Time Frame: Baseline and Week 52 (LOCF)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | New Subjects | Rollover Subjects
Number analyzed (Participants) | 31 | 216
units on a scale | -0.5 (1.3) | -0.5 (1.0)

5. Secondary Outcome: Mean Changes From Baseline in Hamiliton Depression Rating Scale(HAM-D) Item Total Scores at Week 52(LOCF)
Description: The HAM-D was a clinician-rated scale which evaluated the level of depression. The HAM-D consists of 17 items such as depression mood, feeling of guilt, suicide, insomnia, work and activities, retardation, and so on. Each item was scored from 0 to 2, 3 or 4, with higher scores indicating worse condition. Summed subscales were combined to compute a total score. Total score ranges from 0 to 53 , with higher score indicating worse condition.
Time Frame: Baseline and Week 52 (LOCF)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | New Subjects | Rollover Subjects
Number analyzed (Participants) | 31 | 216
units on a scale | -2.2 (8.3) | -4.1 (6.6)

6. Secondary Outcome: Mean Changes From Baseline in Sheehan Disability Scale (SDS) Scores at Week 52(LOCF)
Description: SDS Scale was a patient-rated scale which assessed the degree of impairment for each of 3 items ("work/school," "social life," and "family life/home responsibilities") on a 11-point scale ranging from 0 to 10. The mean SDS score was the mean of scores for 3 items. Higher scores indicate worse condition.
Time Frame: Baseline and Week 52 (LOCF)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | New Subjects | Rollover Subjects
Number analyzed (Participants) | 31 | 216
score on a scale | 0.43 (2.48) | -0.61 (2.35)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from signing of the informed consent form until follow-up for up to 30 days (±5 days) after the final day of IMP administration (end of trial date [final day of observation])
Description: Subjects who received at least one dose of IMP were included in the safety analysis.
Arm/Group | New Subjects | Rollover Subjects
All-Cause Mortality (participants affected / at risk) | 0/31 | 1/216
Serious Adverse Events (participants affected / at risk) | 1/31 | 8/216
Other Adverse Events (participants affected / at risk) | 30/31 | 201/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | New Subjects (N=31) | Rollover Subjects (N=216)
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
HIV infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | New Subjects (N=31) | Rollover Subjects (N=216)
Palpitations (Cardiac disorders) | 3 | 2
Hyperprolactinaemia (Endocrine disorders) | 0 | 11
Hypothyroidism (Endocrine disorders) | 1 | 0
Primary hypogonadism (Endocrine disorders) | 1 | 0
Asthenopia (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 11
Dental caries (Gastrointestinal disorders) | 0 | 7
Dry mouth (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 12
Nausea (Gastrointestinal disorders) | 0 | 12
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 4
Fatigue (General disorders) | 2 | 4
Feeling hot (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 13
Oedema (General disorders) | 1 | 0
Thirst (General disorders) | 2 | 6
Adenoviral conjunctivitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 7
Nasopharyngitis (Infections and infestations) | 5 | 47
Infected dermal cyst (Infections and infestations) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 9
Aspartate aminotransferase increased (Investigations) | 0 | 6
Blood creatine phosphokinase increased (Investigations) | 1 | 4
Blood insulin increased (Investigations) | 0 | 5
Blood prolactin increased (Investigations) | 0 | 9
Blood triglycerides increased (Investigations) | 0 | 8
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 4
Liver function test abnormal (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 7
Weight increased (Investigations) | 4 | 78
Increased appetite (Metabolism and nutrition disorders) | 1 | 17
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Akathisia (Nervous system disorders) | 12 | 46
Bradykinesia (Nervous system disorders) | 3 | 3
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 9
Dyskinesia (Nervous system disorders) | 4 | 7
Dystonia (Nervous system disorders) | 3 | 5
Extrapyramidal disorder (Nervous system disorders) | 4 | 12
Headache (Nervous system disorders) | 1 | 22
Parkinsonism (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 2 | 24
Tremor (Nervous system disorders) | 6 | 15
Anxiety (Psychiatric disorders) | 0 | 5
Depression (Psychiatric disorders) | 1 | 9
Insomnia (Psychiatric disorders) | 2 | 22
Sleep disorder (Psychiatric disorders) | 0 | 8
Major depression (Psychiatric disorders) | 3 | 10
Terminal insomnia (Psychiatric disorders) | 1 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 5
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT03737474/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT03737474/SAP_001.pdf